CLINICAL TRIAL: NCT04729491
Title: Early Antiandrogen Treatment (EAT) With Dutasteride for COVID-19 (EAT-DUTA AndroCoV Trial)
Brief Title: EAT-DUTA AndroCoV Trial
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Corpometria Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CORPO-AB-DRUG-SARS-004B
Record Dates: First submitted 2021-01-25; First posted 2021-01-28 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2020-06

CONDITIONS: Covid19
Keywords: SARS-CoV-2; Dutasteride
MeSH Terms: conditions — COVID-19 | interventions — Dutasteride; Azithromycin; nitazoxanide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dutasteride (Active Comparator): Dutasteride 0.5mg/day q.d. for 30 days or until COVID-19 remission (defined as full remission of symptoms plus viral clearance through rtPCR-SARS-CoV-2)
  Interventions: Drug: Dutasteride 0.5 mg; Drug: Azithromycin; Drug: Nitazoxanide
- Placebo (Placebo Comparator): Placebo q.d. for 30 days or until COVID-19 remission (defined as full remission of symptoms plus viral clearance through rtPCR-SARS-CoV-2)
  Interventions: Drug: Azithromycin; Drug: Nitazoxanide; Drug: Placebo

INTERVENTIONS:
Drug: Dutasteride 0.5 mg — Use of dutasteride 0.5mg/day q.d. for 30 days or until COVID-19 remission, in recently diagnosed COVID-19 subjects.
  Arms: Dutasteride
Drug: Azithromycin — Azithromycin 500mg/day for 05 days
Drug: Nitazoxanide — 500mg twice daily for 06 days
Drug: Placebo — Use of placebo q.d. for 30 days or until COVID-19 remission, in recently diagnosed COVID-19 subjects.
  Arms: Placebo

SUMMARY:
During the continuing SARS-CoV-2 (COVID-19) pandemic, several studies have reported a significant difference in the rate of severe cases between adult females and adult males (42% vs 58%). Among children under the age of 14, the rate of severe cases was reported to be extremely low. To explain this difference, several theories have been proposed including cigarette smoking and lifestyle habits. However, no theory fits both the gender difference in severe cases as well as reduced risk in pre-pubescent children. Our past research on male androgenetic alopecia (AGA) has led us to investigate an association between androgens and COVID-19 pathogenesis. In normal subjects, androgen expression demonstrates significant variation between men and women as well as between adults and pre-pubescent children.

SARS-CoV-2 primarily infects type II pneumocytes in the human lung. SARS-CoV-2 enters pneumocytes, by anchoring to the ACE2 cell surface receptor. Prior to receptor binding, viral spike proteins undergo proteolytic priming by the transmembrane protease, serine 2 (TMPRSS2). TMPRSS2 inhibition or knock down reduces ability of SARS-CoV-1 (a related virus to SARS-CoV-2) to infect cells in vitro. Additionally, TMPRSS2 also facilitates entry of influenza A and influenza B into primary human airway cells and type II pneumocytes.

The human TMPRSS2 gene has a 15 bp androgen response element and in humans, androgens are the only known transcription promoters for the TMPRSS2 gene. In a study of androgen-stimulated prostate cancer cells (LNCaP), TMPRSS2 mRNA expression increase was mediated by the androgen receptor.10 Further, the ACE2 receptor, also critical for SARS-CoV-2 viral infectivity, is affected by male sex hormones with higher activity found in males.

Androgenetic alopecia (AGA), often referred to as male pattern hair loss, is the most common form of hair loss among men. The development of androgenetic alopecia is androgen mediated and is dependent on genetic variants found in the androgen receptor gene located on the X chromosome. We hypothesized that men with AGA would be more prone to severe COVID-19 disease. We conducted a preliminary observational study of hospitalized COVID-19 patients at two Spanish tertiary hospitals between March 23-April 6, 2020 to test this theory. In total, 41 Caucasian males admitted to the hospitals with a diagnosis of bilateral SARS-CoV-2 pneumonia were analyzed. The mean age of patients was 58 years (range 23-79). Among them, 29 (71%) were diagnosed with AGA (16 (39%) were classified as severe AGA (Hamilton IV or above)) and 12 (29%) did not present clinical signs of AGA. The diagnosis of AGA was performed clinically by a dermatologist. The precise prevalence of AGA among otherwise healthy Spanish Caucasian males is unknown; however, based on published literature, the expected prevalence of a similar age-matched Caucasian population is approximately 31-53%.

Further, according to the European Center for Disease Control and Prevention (https://www.ecdc.europa.eu/sites/default/files/documents/covid-19-rapid-risk-assessment-coronavirus-disease-2019-eighth-update-8-april-2020.pdf): "Of the confirmed cases in China, 3.8% (1 716/44 672) were healthcare workers. Of those, 14.8% were severely or critically ill and 5% of the severe cases died. Latest figures reported from Italy show that 9% of COVID-19 cases are healthcare workers, with Lombardy region reporting up to 20% of cases in healthcare workers. In Spain, the latest COVID-19 situation overview from the Ministry of Health reports that 26% of COVID-19 cases are in healthcare workers. In a Dutch study, healthcare workers were tested voluntarily for COVID-19 and 6% tested positive. In a report on 30 cases in healthcare workers in China, all cases had a history of direct contact (distance within 1 metre) with COVID-19 patients, with an average number of 12 contacts, and the average cumulative contact time being two hours (1.5, 2.7). In the Dutch study, only 3% of the healthcare workers reported being exposed to hospital patients with COVID-19 prior onset of symptoms and 63% had worked while asymptomatic.

Based on the scientific rationale combined with this preliminary observation, we propose to test an anti-androgen as a treatment for patients recently diagnosed with COVID-19. This study is intended to explore the possible protective role of anti-androgens in SARS-CoV-2 infection, including reduction of virological duration and disease severity.

ELIGIBILITY:
Inclusion Criteria:

1. Male
2. ≥18 years old
3. Laboratory confirmed positive SARS-CoV-2 rtPCR test within 7 days prior to randomization
4. Clinical status on the COVID-19 Ordinal Scale (defined in Section 5.1) of 1 to 3
5. Subject (or legally authorized representative) gives written informed consent prior to performing any study procedures
6. Subject (or legally authorized representative) agree that subject will not participate in another COVID-19 trial while participating in this study

Exclusion Criteria:

1. Subject enrolled in a study to investigate a treatment for COVID-19
2. Require oxygen use, hospitalization or mechanical ventilation
3. Tachycardia (HR > 150 bpm) or hypotension (BP < 90/60 mmHg)
4. Patients who are allergic to the investigational product or similar drugs (or any excipients);
5. Subjects with QTcF > 450 ms
6. Subjects with uncontrolled medical conditions that could compromise participation in the study - uncontrolled hypertension (BP > 220/120 mmHg), uncontrolled hypothyroidism (TSH > 10 iU/L), uncontrolled diabetes mellitus (HbA1c > 12%)
7. Alanine Transaminase (ALT) or Aspartate Transaminase (AST) > 5 times the upper limit of normal.
8. Estimated glomerular filtration rate (eGFR) < 30 ml/min or requiring dialysis
9. Subject (or legally authorized representative) not willing or unable to provide informed consent
10. Not willing to provide informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-10-07 (Actual)

PRIMARY OUTCOMES:
Positivity rate of rtPCR-SARS-CoV-2 (qualitative analysis) | Day 7
  Treatment efficacy of dutasteride relative to placebo arm as assessed by viral load measured by positivity rate (% of positive, detected rtSARS-CoV-2)

SECONDARY OUTCOMES:
World Health Organization (WHO) Clinical Progression Scale [0 to 10; 0 = uninfected; 10 = death] | Day 14
  Treatment efficacy of dutasteride relative to placebo arm as assessed by World Health Organization (WHO) Clinical Progression Scale [0 to 10; 0 = uninfected; 10 = death]
World Health Organization (WHO) COVID=19 Ordinal Scale for Clinical Improvement [1 to 8; 1 = not hospitalized, no limitation on activities; 8 = death] | Day 7
  Treatment efficacy of dutasteride relative to placebo arm as assessed by World Health Organization (WHO) COVID=19 Ordinal Scale for Clinical Improvement [1 to 8; 1 = not hospitalized, no limitation on activities; 8 = death]
Time-to-recovery | Day 28
  Recovery is defined as the first day on which the subject satisfies category one from the COVID ordinal scale (defined in Section 5.1): (1) Not hospitalized, no limitations on activities. [Parameter: Number of days until achieve Category 1 of the World Health Organization (WHO) COVID=19 Ordinal Scale for Clinical Improvement [1 to 8; 1 = not hospitalized, no limitation on activities; 8 = death]
SARS-CoV-2 viral load | Day 5
  Treatment efficacy dutasteride relative to placebo arm as assessed by viral load measured by rtPCR-SARS-CoV-2 (CTs)
Duration of fatigue | Day 14
  Treatment efficacy of dutasteride relative to placebo arm as assessed by duration of fatigue (days)
Duration of anosmia | Day 14
  Treatment efficacy of dutasteride relative to placebo arm as assessed by duration of anosmia (days)
Overall duration of clinical manifestations | Day 14
  Treatment efficacy of dutasteride relative to placebo arm as assessed by duration of overall symptoms (days)
Proportion of subjects needing additional drugs or interventions | Day 28
  Defined as the number of subjects who have required additional drugs (glucocorticoids, anticoagulants, etc) or interventions allocated to each arm divided by the number of subjects randomized to that specific arm (%). Treatment efficacy dutasteride relative to placebo arm as assessed by the proportion of subjects needing additional drugs or interventions in each arm. (%)
Proportion of subjects needing oxygen use | Day 28
  Defined as the number of subjects who have required oxygen use allocated to each arm divided by the number of subjects randomized to that specific arm (%). Treatment efficacy of dutasteride relative to placebo arm as assessed by the proportion of subjects needing oxygen use in each arm. (%)
Proportion of subjects needing high-flow oxygen therapy or non-invasive ventilation | Day 28
  Defined as the number of subjects who have required high-flow oxygen use or non-invasive mechanical ventilation allocated to each arm divided by the number of subjects randomized to that specific arm (%). Treatment efficacy of dutasteride relative to placebo arm as assessed by the proportion of subjects needing high-flow oxygen use or non-invasive mechanical ventilation in each arm.
Proportion of hospitalizations | Day 28
  Defined as the number of hospitalizations in each arm divided by the number of subjects randomized to that specific arm (%). Treatment efficacy of dutasteride relative to placebo arm as assessed by the proportion of hospitalizations in each arm.
Proportion of mechanical ventilation use | Day 28
  Defined as the number of subjects that needed mechanical ventilation in each arm divided by the number of subjects randomized to that specific arm (%). Treatment efficacy of dutasteride relative to placebo arm as assessed by the number of mechanical ventilation use in each arm divided by the number of subjects randomized to that specific arm.
Proportion of vasopressors use | Day 28
  Defined as the number of subjects that needed vasopressors use in each arm divided by the number of subjects randomized to that specific arm (%).Treatment efficacy of dutasteride relative to placebo arm as assessed by the number of subjects needing use of pressors in each arm divided by the number of subjects randomized to that specific arm.
Proportion of deaths | Day 60
  Treatment efficacy of dutasteride relative to placebo arm as assessed by the number of subjects who have died in each arm divided by the numbers of subjects randomized to the treatment arm (%).
Duration of new oxygen use | Day 28
  Treatment efficacy of dutasteride relative to placebo arm as assessed by the duration of new oxygen use measured in days among subjects that did not require oxygen upon randomization and required oxygen use after the beginning of treatment, in each arm (days)
Duration of hospitalization | Day 28
  Treatment efficacy of dutasteride relative to placebo arm as assessed by the duration of hospitalization measured in days among subjects that required hospitalization, in each arm (days)
Duration of mechanical ventilation | Day 28
  Treatment efficacy of dutasteride relative to placebo arm as assessed by the duration of mechanical ventilation measured in days among subjects that required mechanical ventilation, in each arm (days)
Proportion of increased ultrasensitive C-reactive protein (usCRP) (defined as usRCP > 7 mg/L) | Day 1
  Treatment efficacy of dutasteride relative to placebo arm as assessed by the number of subjects presenting increased ultrasensitive C-reactive protein (usCRP) at Day 1, divided by the number of subjects randomized to that specific arm (%).
Proportion of increased ultrasensitive C-reactive protein (usCRP) (defined as usRCP > 7 mg/L) | Day 3
  Treatment efficacy of dutasteride relative to placebo arm as assessed by the number of subjects presenting increased ultrasensitive C-reactive protein (usCRP) at Day 3, divided by the number of subjects randomized to that specific arm (%).
Proportion of increased ultrasensitive C-reactive protein (usCRP) (defined as usRCP > 7 mg/L) | Day 7
  Treatment efficacy of dutasteride relative to placebo arm as assessed by the number of subjects presenting increased ultrasensitive C-reactive protein (usCRP) at Day 7, divided by the number of subjects randomized to that specific arm (%).
Proportion of decrease in erythrocyte sedimentation rate (ESR) (defined as ESR decrease > 50% compared to baseline (Day 0)) | Day 1
  Treatment efficacy of dutasteride relative to placebo arm as assessed by the number of subjects presenting ESR decrease > 50% at Day 1, divided by the number of subjects randomized to that specific arm (%).
Proportion of decrease in erythrocyte sedimentation rate (ESR) (defined as ESR decrease > 50% compared to baseline (Day 0)) | Day 3
  Treatment efficacy of dutasteride relative to placebo arm as assessed by the number of subjects presenting ESR decrease > 50% at Day 3, divided by the number of subjects randomized to that specific arm (%).
Proportion of decrease in erythrocyte sedimentation rate (ESR) (defined as ESR decrease > 50% compared to baseline (Day 0)) | Day 7
  Treatment efficacy of dutasteride relative to placebo arm as assessed by the number of subjects presenting ESR decrease > 50% at Day 7, divided by the number of subjects randomized to that specific arm (%).
Proportion of increase in eosinophils (defined as eosinophils increase > 50% compared to baseline (Day 0)) | Day 1
  Treatment efficacy of dutasteride relative to placebo arm as assessed by the number of subjects presenting eosinophils increase > 50% at Day 1, divided by the number of subjects randomized to that specific arm (%).
Proportion of increase in eosinophils (defined as eosinophils increase > 50% compared to baseline (Day 0)) | Day 3
  Treatment efficacy of dutasteride relative to placebo arm as assessed by the number of subjects presenting eosinophils increase > 50% at Day 3, divided by the number of subjects randomized to that specific arm (%).
Proportion of increase in eosinophils (defined as eosinophils increase > 50% compared to baseline (Day 0)) | Day 7
  Treatment efficacy of dutasteride relative to placebo arm as assessed by the number of subjects presenting eosinophils increase > 50% at Day 7, divided by the number of subjects randomized to that specific arm (%).
Proportion of increased d-dimer (defined as d-dimer > 500 mg/dL) | Day 7
  Treatment efficacy of dutasteride relative to placebo arm as assessed by the number of subjects presenting increased d-dimer protein (usCRP) at Day 7, divided by the number of subjects randomized to that specific arm (%).
Variation in oxygen saturation compared to baseline (Day 0) | Day 1
  Treatment efficacy of dutasteride relative to placebo arm as assessed by the mean variation of oxygen saturation of subjects randomized to that specific arm (%) at Day 1 compared to baseline (Day 0).
Variation in oxygen saturation compared to baseline (Day 0) | Day 3
  Treatment efficacy of dutasteride relative to placebo arm as assessed by the mean variation of oxygen saturation of subjects randomized to that specific arm (%) at Day 3 compared to baseline (Day 0).
Variation in oxygen saturation compared to baseline (Day 0) | Day 5
  Treatment efficacy of dutasteride relative to placebo arm as assessed by the mean variation of oxygen saturation of subjects randomized to that specific arm (%) at Day 5 compared to baseline (Day 0).
Variation in oxygen saturation compared to baseline (Day 0) | Day 7
  Treatment efficacy of dutasteride relative to placebo arm as assessed by the mean variation of oxygen saturation of subjects randomized to that specific arm (%) at Day 7 compared to baseline (Day 0).
Disease duration | Day 30
  Treatment efficacy of dutasteride relative to placebo arm as assessed by duration of symptoms, complications, or any other COVID-related clinical or biochemical sign of disease (days)
Change in viral load from baseline to Day 5 | Day 5
  Treatment efficacy of dutasteride relative to placebo arm as assessed by change in viral load from baseline to Day 5 measured by rtPCR-SARS-CoV-2 (CTs)
Proportion of post-COVID mental symptoms | Day 30
  Treatment efficacy of dutasteride relative to placebo arm as assessed by the number of subjects persisting with mental symptoms after COVID-19 resolution in each arm divided by the number of subjects randomized to that specific arm (%) at Day 30.
Proportion of post-COVID physical symptoms | Day 30
  Treatment efficacy of dutasteride relative to placebo arm as assessed by the number of subjects persisting with physical symptoms after COVID-19 resolution in each arm divided by the number of subjects randomized to that specific arm (%) at Day 30.
Proportion of post-COVID overall symptoms | Day 30
  Treatment efficacy of dutasteride relative to placebo arm as assessed by the number of subjects persisting with any symptoms after COVID-19 resolution in each arm divided by the number of subjects randomized to that specific arm (%) at Day 30.
Proportion of post-COVID mental symptoms | Day 60
  Treatment efficacy of dutasteride relative to placebo arm as assessed by the number of subjects persisting with mental symptoms after COVID-19 resolution in each arm divided by the number of subjects randomized to that specific arm (%) at Day 60.
Proportion of post-COVID physical symptoms | Day 60
  Treatment efficacy of dutasteride relative to placebo arm as assessed by the number of subjects persisting with physical symptoms after COVID-19 resolution in each arm divided by the number of subjects randomized to that specific arm (%) at Day 60.
Proportion of post-COVID overall symptoms | Day 60
  Treatment efficacy of dutasteride relative to placebo arm as assessed by the number of subjects persisting with any symptoms after COVID-19 resolution in each arm divided by the number of subjects randomized to that specific arm (%) at Day 60.
Proportion of post-COVID mental symptoms | Day 90
  Treatment efficacy of dutasteride relative to placebo arm as assessed by the number of subjects persisting with mental symptoms after COVID-19 resolution in each arm divided by the number of subjects randomized to that specific arm (%) at Day 90.
Proportion of post-COVID physical symptoms | Day 90
  Treatment efficacy of dutasteride relative to placebo arm as assessed by the number of subjects persisting with physical symptoms after COVID-19 resolution in each arm divided by the number of subjects randomized to that specific arm (%) at Day 90.
Proportion of post-COVID overall symptoms | Day 90
  Treatment efficacy of dutasteride relative to placebo arm as assessed by the number of subjects persisting with any symptoms after COVID-19 resolution in each arm divided by the number of subjects randomized to that specific arm (%) at Day 90.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos G. Wambier, MD, Ph.D., Study Director — Alpert School of Medicine - Brown University; Flavio A. Cadegiani, MD, MSc, Ph.D., Principal Investigator — Corpometria Institute; Andy Goren, MD, Study Chair — Applied Biology
Locations (1):
- Corpometria Institute, Brasília, Federal District, Brazil

IPD SHARING:
Plan to Share IPD: No